CLINICAL TRIAL: NCT00377351
Title: Confirmation of Self-Reported Incident ALS Cases in the AARP-Diet and Health (AARP-DH) Cohort
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906247; 06-E-N247
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Public Health; Elderly Population; Neurodegenerative Diseases; Exposure; Lifestyle
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Neurodegenerative Diseases

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a rare but rapidly progressive neurological disease that often results in death within a few years after the diagnosis. The incidence of ALS in the US is approximately 2.0/100,000/year and is age dependent. Very few epidemiological studies have investigated the causes of ALS. Last year, Dr. Alberto Ascherio at Harvard School of Public Health successfully obtained a RO1 grant to investigate the risk of ALS by documenting ALS cases in five well-established large prospective cohorts: The Nurses' Health Study (NHS), the Health Professionals Follow-up Study (HPFS), the Cancer Prevention Study II Nutrition Cohort (CPS IIN), the Multiethnic Cohort (MEC), and the NIH-American Association of Retired Persons Diet and Health Study (AARP-DH). The primary aims of this grant are to prospectively clarify the associations between diet and smoking and risk of ALS in this to date the largest epidemiological study on ALS. Incident ALS cases will be documented via biennial questionnaires in the first three cohorts. While mortality data will be obtained in the MEC and AARP-DH cohorts by searching the National Death Index (NDI) Plus, it is also desirable to identify surviving incident cases in these two cohorts.

The objective of this specific proposal is to ascertain the self-reported incident ALS cases from the AARP-DH study and obtain consent for medical release following the procedures set up for Parkinson's disease (PD) cases in the currently approved Parkinson's Genes and Environment (PAGE) Study IRB approval #06-E-N093. The confirmed ALS cases may be analyzed as part of the RO1 project. We expect to identify 300 self-reported ALS cases from the AARP cohort. Detailed analytic plans will be coordinated with Dr. Ascherio.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a rare but rapidly progressive neurological disease that often results in death within a few years after the diagnosis. The incidence of ALS in the US is approximately 2.0/100,000/year and is age dependent. Very few epidemiological studies have investigated the causes of ALS. Last year, Dr. Alberto Ascherio at Harvard School of Public Health successfully obtained a RO1 grant to investigate the risk of ALS by documenting ALS cases in five well-established large prospective cohorts: The Nurses' Health Study (NHS), the Health Professionals Follow-up Study (HPFS), the Cancer Prevention Study II Nutrition Cohort (CPS IIN), the Multiethnic Cohort (MEC), and the NIH-American Association of Retired Persons Diet and Health Study (AARP-DH). The primary aims of this grant are to prospectively clarify the associations between diet and smoking and risk of ALS in this to date the largest epidemiological study on ALS. Incident ALS cases will be documented via biennial questionnaires in the first three cohorts. While mortality data will be obtained in the MEC and AARP-DH cohorts by searching the National Death Index (NDI) Plus, it is also desirable to identify surviving incident cases in these two cohorts.

The objective of this specific proposal is to ascertain the self-reported incident ALS cases from the AARP-DH study and obtain consent for medical release following the procedures set up for Parkinson's disease (PD) cases in the currently approved Parkinson's Genes and Environment (PAGE) Study IRB approval #06-E-N093. The confirmed ALS cases may be analyzed as part of the RO1 project. We expect to identify 300 self-reported ALS cases from the AARP cohort. Detailed analytic plans will be coordinated with Dr. Ascherio.

ELIGIBILITY:
* INCLUSION CRITERIA:

This study will be conducted within the infrastructure of the NIH-AARP Diet and Health Study; every participant in the AARP cohort self-reporting an ALS diagnosis will be eligible for the current investigation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-09-11; Study Completion 2010-08-03

CONTACTS AND LOCATIONS:
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] McGuire V, Longstreth WT Jr, Koepsell TD, van Belle G. Incidence of amyotrophic lateral sclerosis in three counties in western Washington state. Neurology. 1996 Aug;47(2):571-3. doi: 10.1212/wnl.47.2.571. PMID 8757041
- [Background] Kamel F, Umbach DM, Lehman TA, Park LP, Munsat TL, Shefner JM, Sandler DP, Hu H, Taylor JA. Amyotrophic lateral sclerosis, lead, and genetic susceptibility: polymorphisms in the delta-aminolevulinic acid dehydratase and vitamin D receptor genes. Environ Health Perspect. 2003 Aug;111(10):1335-9. doi: 10.1289/ehp.6109. PMID 12896855
- [Background] Kamel F, Umbach DM, Munsat TL, Shefner JM, Hu H, Sandler DP. Lead exposure and amyotrophic lateral sclerosis. Epidemiology. 2002 May;13(3):311-9. doi: 10.1097/00001648-200205000-00012. PMID 11964933